CLINICAL TRIAL: NCT00472927
Title: An Open-Label, Single-Dose, Randomized, 4-Period, Crossover, Bioequivalence Study of Three New Formulations of Premarin 0.45mg/Medroxyprogesterone Acetate (MPA) 1.5mg Compared With a Reference Formulation of Premarin/MPA (PremproTM) 0.45mg/1.5mg in Healthy Postmenopausal Women
Brief Title: Bioequivalence Study of 3 New Formulations of Premarin/MPA Compared With Premarin/MPA (Prempro)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0713E1-1142
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Postmenopause

INTERVENTIONS:
Drug: Premarin/MPA 0.45 mg/1.5 mg

SUMMARY:
To evaluate three new investigational tablet formulations of the Food and Drug Administration (FDA) approved medication Prempro™, Premarin combined with medroxyprogesterone acetate (MPA).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, postmenopausal women, aged 35 to 70 years
* Spontaneous amenorrhea for at least 12 months (no FSH required) or spontaneous amenorrhea for at least 6 months (FSH level ≥38 mIU/mL); spontaneous amenorrhea must have begun by the age of 55
* BMI in the range of 18 to 35 kg/m2

Exclusion Criteria:

* History or presence of hypertension (>139 mm Hg systolic or >89 mm Hg diastolic)
* History of drug allergy to conjugated estrogens (CE) or selective estrogen receptor modulators (SERMs)
* Use of prescription or investigatioanl drugs within 30 days before test article administration

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-05; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentration data and PK parameters of MPA and Premarin (esrone and equilin components)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Miami, Florida, United States